CLINICAL TRIAL: NCT05155930
Title: Evaluation of the Efficacy of Internal Family Systems (IFS) Therapy for Trauma-related Symptoms Among Complexly Traumatized Adults
Brief Title: Evaluation of the Efficacy of Internal Family Systems (IFS) Therapy
Acronym: IFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justice Resource Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JRI 2014-02
Record Dates: First submitted 2017-03-24; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: PTSD; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: The Internal Family Systems (IFS) model of psychotherapy is a trauma-informed promising practice that has shown promise for individuals who struggle with trauma related symptoms including PTSD, dissociation and depression, as well as disruptions in self-concept and self-regulation. IFS places a heavy emphasis on aiding individuals in building an internalized sense of self-efficacy and self-compassion that may then support the development of self-regulatory capacity and reductions in trauma-related symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IFS (Experimental): Internal Family Systems (IFS)
  Interventions: Behavioral: Internal Family Systems (IFS)

INTERVENTIONS:
Behavioral: Internal Family Systems (IFS) — Weekly individual psychotherapy

SUMMARY:
Study examining the effectiveness of 16 weeks of Internal Family Systems (IFS) therapy for adults with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Evaluation study of IFS therapy among trauma-impacted adults in order to explore the applicability of IFS with this population, ensure fidelity of treatment administration, and examine initial efficacy. Evaluate the utility of IFS in reducing symptoms of PTSD, dissociation and depression and increasing self-regulatory capacity, self-awareness and self-compassion. 15 subjects between the ages of 18 and 56 who are receiving 16, 90-minute sessions of IFS therapy by certified IFS practitioners in the community will be recruited for this evaluation study. Blind evaluators will assess treatment effects at pre-treatment, mid-treatment, post-treatment and at one-month follow-up, measuring change in symptoms of PTSD, dissociation and depression, as well as self-regulation, self-compassion, and interoceptive awareness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 58 years old, any race.
* A minimum two traumatic events prior to the age of 18 years.
* Current PTSD diagnosis per CAPS assessment with total symptom scores indicative of a moderate degree of severity (i.e. CAPS total score between 55 and 80).
* Clinically significant depressive symptoms as indicated by a total score of 14 or above on the BDI.

Exclusion Criteria:

* GAF < 40.
* Diagnosis of schizophrenia, DID, Bipolar Disorder or other psychotic disorder not stated above.
* Substance dependence or abuse in the past 6 months, as defined by DSM IV criteria and judged by the PI.
* Current legal proceedings resulting from the traumatic events.
* Previous treatment in IFS.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS) total score from pre- to post-treatment and 1-month follow up | Change from baseline in PTSD symptom severity at up to 16 weeks of treatment and 1-month follow up.
  A 30-item validated instrument that contains frequency and intensity scales for PTSD symptoms . Subscales assess intrusion, avoidance, arousal and associated affective features.

SECONDARY OUTCOMES:
Change in PTSD symptoms per the Davidson Trauma Scale (DTS) across four study time points | Change from baseline in PTSD symptom severity at up to 8 weeks of treatment, 16 weeks of treatment and 1-month follow up.
  Self-report of PTSD symptoms per DSM IV criteria.
Change in symptoms of depression per the Beck Depression Inventory (BDI) across 4 study time points | Change from baseline in PTSD symptom severity at up to 8 weeks of treatment, 16 weeks of treatment and 1-month follow up.
  21-item, self-report measure of symptoms of depression.
Change in interoceptive awareness per the Multidimensional Assessment of Interoceptive Awareness (MAIA) across 4 study time points | Change from baseline in PTSD symptom severity at up to 8 weeks of treatment, 16 weeks of treatment and 1-month follow up.
  32-item, self-report measure that assesses interoceptive body awareness across eight distinct but related dimensions: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting.
Change in symptoms of dissociation per the Structured Interview for Disorders of Extreme Stress, Self-Report Version (SIDES-SR) over 4 study time points | Change from baseline in PTSD symptom severity at up to 8 weeks of treatment, 16 weeks of treatment and 1-month follow up.
  45 item, validated self-report measure assessing six domains of impairment secondary to complex trauma exposure. Assessed areas include alterations in (a) regulation of affect and impulses, (b) attention and consciousness, (c) self-perception, (d) relation with others, (e) somatization, and (f) systems of meaning.
Change in self-compassion per the Self Compassion Scale over four study time points | Change from baseline in PTSD symptom severity at up to 8 weeks of treatment, 16 weeks of treatment and 1-month follow up.
  26 item self report outcome measure assessing components of compassion towards the self including self-kindness, common humanity, and mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Hodgdon, Ph.D., Principal Investigator — Trauma Center

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Hodgdon, H.B., Gustella-Anderson, F., Southwell, E., Hrubec, W., & Schwartz, R. (November, 2017). Pilot Study of Internal Family Systems Therapy for Adults with a History of Childhood Trauma and Chronic PTSD. Poster presented at the annual meeting of International Society of Traumatic Stress Studies (ISTSS),Chicago, IL.